CLINICAL TRIAL: NCT01668160
Title: Analysis of the Stability of Total Hip Arthroplasty Implants Used in Revision Surgery Using Radiostereometric Analysis (RSA)
Brief Title: Stability of Revision Total Hip Arthroplasty Implants Using Radiostereometric Analysis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Charles R. Bragdon, Reseach scientist, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012P000925; 216494 (Other Grant/Funding Number: MGH Orhtopaedic Department Funds 216494)
Record Dates: First submitted 2012-08-10; First posted 2012-08-17 (Estimated); Last update posted 2013-11-05 (Estimated); Status verified 2013-11

CONDITIONS: Osteoarthritis of Hip; Failure of Primary THA
Keywords: clinical outcomes; radiographic outcomes; total hip arthroplasty; survivorship
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Revision Total Hip (Experimental): patients recieving a revision total hip replacement will be assessed for implant stability and wear using RSA. Tantalum beads will be placed in the polyethylene and surrounding pelvic and femoral bone.
  Interventions: Procedure: Bead placement during revision hip replacement surgery

INTERVENTIONS:
Procedure: Bead placement during revision hip replacement surgery — Tantalum beads will be placed in the surrounding pelvic and femoral bone and the polyethylene component during surgical treatment of failed primary THA components

SUMMARY:
The specific aim is to quantify the stability of the acetabular and femoral components of a revision total hip arthroplasty (THA) in vivo as currently performed at our institution. In this way, the investigators will gain insight into the outcome of the current state of the art of revision arthroplasty surgery. In the past, acetabular and femoral component stability has been measured using radiostereometric analysis (RSA) and when patients having revision total hip operations were compared to patients undergoing primary total hip operations it was possible to determine differences in stability and this was predictive of the intermediate to long-term performance of the acetabular and femoral reconstruction. The investigators propose to use this established, high resolution technique to assess and compare the stability of the revision implants.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female.
2. 25 to 75 years of age.
3. Subjects requiring revision total hip replacement.
4. Subjects who demonstrate the ability to return to MGH for follow-up for the next five years.

Exclusion Criteria:

1. Subjects with limited life span.
2. Subjects with difficulty in comprehending study protocol for any reason.
3. Subjects with complex disease entities which significantly increase the risks of the surgery such as any major platelet abnormality, hematological disorder, or any other major medical complication which could substantially reduce longevity, put them at further risk due to immunocompromisation or increase the risk of infection.
4. Female subjects that are pregnant or who may suspect they are pregnant or who plan to become pregnant while participating in this study.

   * A urine HCG will be done in all women of child bearing potential prior to RSA imaging at each follow-up visit. The result will be recorded in the research record.

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-02; Primary Completion 2020-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Stability of Acetabular and femoral components | 1, 2, 3, 5 years after surgery
  RSA films will be taken at the prescribed time intervals to measure component mothion over time.

SECONDARY OUTCOMES:
Wear of the polyethlene component | 1, 2, 3, 5 years after surgery
  The movement of the femoral head into the polyethylenen, (wear), will be measured at the prescribed time intervals.

OTHER OUTCOMES:
Assessment/questionaire HOOS | Pre-op, 1, 2, 3, 5 years after surgery
  Hip disability and Osteoarthritis Outcome Score
Assessment/Questionaires Harris Hip Score | Pre-op, 1, 2, 3, 5 years after surgery
  Hip specific questionaire
Assessment/Questionaire UCLA Activity Score | Pre-op, 1, 2, 3, 5 years after surgery
  Measure of activity level
Assessment/Questionaire EQ-5D | Pre-op, 1, 2, 3, 5 years after surgery
  General health and cost effectiveness measure
Assessment/Questionaire Case Mix indicator | Pre-op, 1, 3, 5, 7, 10 years after surgery
  Determines comorbidities

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States